CLINICAL TRIAL: NCT01166477
Title: Ensayo clínico, Abierto, Aleatorizado Para Comparar la Calidad de Vida de Los Pacientes VIH+ Que Inician Monoterapia Con Comprimidos de LPV/r vs Triple Terapia Que Contenga un IP Potenciado
Brief Title: Clinical Trial, Open-label, Randomised, in Order to Compare the Quality of Life for Those VIH+ Patients That Start With Monotherapy on LPV/r Tablets Vs. Triple Therapy With a Boosted Protease Inhibitor
Acronym: QoLKAMON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sociedad Andaluza de Enfermedades Infecciosas (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAI-CDV-2009-01
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2009-10

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — lopinavir-ritonavir drug combination; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triple therapy (Active Comparator): The patients who would be allocated to this arm will continue with their triple therapy treatment, based on any protease inhibitor boosted with ritonavir
  Interventions: Drug: Triple therapy with ritonavir
- Monotherapy (Experimental): Those patients allocated to this arm will start to take Kaletra (lopinavir200mg/ritonavir50mg)two tablets bid
  Interventions: Drug: Lopinavir and ritonavir

INTERVENTIONS:
Drug: Lopinavir and ritonavir — The patients will take Kaletra (lopinavir200mg/ritonavir50mg)two tablets bid
  Arms: Monotherapy
Drug: Triple therapy with ritonavir — The patients will continue to take their usual triple therapy, as established in the summary of product characteristics
  Arms: Triple therapy

SUMMARY:
The Study will help to compare the Quality of Life for those HIV patients that are on monotherapy with LPV/r Vs. triple therapy with a boosted protease inhibitor

DETAILED DESCRIPTION:
The Study will help to compare the Quality of Life for those HIV patients that are on monotherapy with LPV/r Vs. triple therapy with a boosted protease inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with HIV-1, documented with a positive HIV-1 antibodies test and/or positive PCR confirmed for HIV-1 RNA.
* Patients on triple antiretroviral therapy with any boosted protease inhibitor.
* Patients with an undetectable viral load, which will be defined as <50 viral RNA copies/mL within the last six months.
* Men or women aged≥18.
* For women with childbearing potential, negative urine pregnancy test during the Screening visit.
* Patients who would have granted a written informed consent prior to any Study-specific screening procedure.

Exclusion Criteria:

* Patients with a written proof of resistance in the accumulated genotype, which would lead to a sensibility loss to lopinavir/ritonavir, or, in case of genotype absence, a documented failure to a protease inhibitor therapy.
* Patients with a CD4 cells nadir CD4 <100 cell/microL.
* Patients who, for any reason, could not be treated with lopinavir/ritonavir.
* Prior medical history of psychiatric disorders, such as depressive syndrome, schizophrenia or psychotic disease.
* Known previous medical history of drug abuse/addiction or alcohol chronic consumption, which in the Investigator's opinion, would be incompatible with his/her Study participation.
* Pregnant or breastfeeding women, or women of childbearing potential who do not use an appropriate contraceptive method, according to the Investigator's opinion.
* Documented past(within four weeks prior to screening) or active current opportunistic infection.
* Patients who, due to severe toxicities related to any of their current HAART compounds, there is a planned discontinuation or modification concerning any of the drugs from their triple therapy.
* Patients for which, according to the Investigator, will have to change their HAART, regardless of the reason, within the next six months.
* Renal disease with creatinine clearance <60 mL/min.
* Concomitant use of Lopinavir/ritonavir contraindicated drugs, such as rifampicin, dihydroergotamine, ergotamine, methylergonovine, cisapride, hypericum perforatum, lovastatin, simvastatin, pimozide, midazolam and triazolam.
* Concomitant use of nephrotoxic or immunosuppressor drugs.
* Patients currently treated with systemic corticosteroids, interleukine-2 or chemotherapy.
* Patients treated with other Investigative Medical Product.
* Patients with acute hepatitis.
* Any disease or condition that, according to the Investigator, would be incompatible with the patient's participation in the Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Quality of Life comparison for HIV patients that start monotherapy with lopinavir/ritonavir (LPV/r) tablets vs patients with triple therapy which would include any boosted protease inhibitor (PI). | 24 weeks per patients

SECONDARY OUTCOMES:
Virologic efficacy assessment for HIV patients on monotherapy based on LPV/r tablet vs triple therapy which would include any protease inhibitor | 24 weeks per patient
Immune response changes assessment for those HIV patients who start monotherapy with LPV/r tablets vs HIV patients on triple therapy which would include any protease inhibitor | 24 weeks per patients
Patient satisfaction assessment for HIV patients that start monotherapy with LPV/r tablets vs triple therapy which would include any protease inhibitor | 24 weeks per patient
Treatment adherence assessment for HIV patients who start on LPV/r monotherapy tablets vs triple therapy which include any protease inhibitor | 24 weeks per patient
Tolerability and safety assessment for the HIV patients who start monotherapy treatment with LPV/r tablets vs triple therapy which would include any protease inhibitor | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pasquau, MD, Principal Investigator — Sociedad Andaluza de Enfermedades Infecciosas
Locations (31):
- Spain (31):
  - Hospital de San Juan, San Juan, Alicante
  - Hospital de Torrevieja, Torrevieja, Alicante
  - Hospital de Villajoyosa, Villajoyosa, Alicante
  - Hospital de Torrecárdenas, Almería, Almería
  - Hospital General de l'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Yagüe, Burgos, Burgos
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Hospital Puerto Real, Cadiz, Cádiz
  - Hospital Clínico San Cecilio, Granada, Granada
  - Hospital Virgen de las Nieves, Granada, Granada
  - Pilar Vázquez Rodríguez, A Coruña, La Coruña
  - Hospital Clínico Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Carlos Haya, Málaga, Málaga
  - Hospital Clínico de Málaga, Málaga, Málaga
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Hospital de Valme, Seville, Sevilla
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Virgen de la Cinta, Tortosa, Tarragona
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital de Basurto, Basurto, Vizcaya
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza